CLINICAL TRIAL: NCT01935583
Title: Intervention to Promote Survivor Resilience and Adjustment: Efficacy Evaluation (a Research Project Within the Traumatic Brain Injury Model System Grant)
Brief Title: Intervention to Promote Survivor Resilience and Adjustment: Efficacy Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM14738; H133A120031 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2013-08-21; First posted 2013-09-05 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resilience/Adjustment Counseling (Experimental): Intervention to promote resilience and adjustment (RAI) - The RAI was developed based upon considerable clinical experience and research review. The RAI is a structured approach to helping individuals after brain injury address issues related to resilience and adjustment to injury. The RAI is implemented in seven, 60-minute, in-person sessions.
  Interventions: Behavioral: Resilience/Adjustment Counseling
- Waitlist Control (No Intervention): Individuals are randomly assigned to the treatment group or waitlist control (WLC) group. Individuals will complete the study measures on 2 occasions, 5 weeks apart. In fairness, WLC participants will then be offered the opportunity to participate in the intervention.

INTERVENTIONS:
Behavioral: Resilience/Adjustment Counseling — Intervention to promote individual's resilience and adjustment (RAI) - The RAI is a structured approach to helping individuals after brain injury address issues related to resilience and adjustment. The RAI is implemented in seven sessions. Each session is in-person and lasts for 60 minutes.
  Arms: Resilience/Adjustment Counseling

SUMMARY:
1. To evaluate the short and longer-term efficacy of a structured outpatient intervention program (The Resilience and Adjustment Intervention, RAI) to improve survivors' resilience.
2. To evaluate the impact of treatment on emotional well-being and postinjury adjustment.
3. To evaluate the impact of the intervention on abilities including problem solving, communication, and stress management.
4. To examine the extent to which treatment benefits are sustained in the longer-term.

DETAILED DESCRIPTION:
To design effective resilience interventions, a treatment modality which is effective for traumatic brain injury (TBI) survivors is needed. Virginia Commonwealth University (VCU) researchers have had considerable success in the past several decades developing and evaluating interventions for neurobehavioral, cognitive, and vocational challenges after TBI. Researchers have demonstrated the utility of the curriculum-based (C-B) treatment structure in various settings. Additionally, the efficacy of the C-B structure, independent of postinjury timeframe, allows the flexibility necessary to address the unique consequences of TBI.

The C-B treatment modality offers a promising strategy for the promotion of resilience postinjury. The primary purpose of the study is to evaluate the efficacy of a structured, curriculum-based intervention to promote postinjury resilience and adjustment. Objectives include:

1. to evaluate the short and longer-term efficacy of a structured outpatient intervention program (The Resilience and Adjustment Intervention, RAI) to improve survivors' resilience
2. to evaluate the impact of treatment on emotional well-being and postinjury adjustment
3. to evaluate the impact of the intervention on abilities including problem solving, communication, and stress management
4. to examine the extent to which treatment benefits are sustained in the longer-term

ELIGIBILITY:
Inclusion Criteria:

* mild, moderate, or severe TBI
* able to understand and provide consent

Exclusion Criteria:

* active substance abusers (e.g., intoxicated at arrival to intake)
* at imminent risk of psychiatric hospitalization
* in imminent danger of hurting themselves or others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2013-01; Primary Completion 2016-10 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Connor-Davidson Resilience Scale-10 (CD-RISC-10) | Change from Baseline to Post-Treatment (5 weeks after Baseline)
  During the past decade, researchers have developed resilience measurement scales, and a recent review suggested that Connor and Davidson have been most successful. The authors first developed a 25 item scale (CD-RISC) reflecting resilience characteristics identified by Kobasa and Rutter. Normative studies including factor analyses indicated that the CD-RISC is reliable, valid, and sensitive to treatment effects. More recently, a 10-item version was developed using exploratory and confirmatory factors analyses. Respondents are presented with a series of descriptors (e.g., "I am able to adapt and change," "Coping with stress can strengthen me") and rate themselves on a 0 - 4 scale ranging from rarely true (0) to true nearly all the time (4). Campbell-Sills and colleagues have characterized the 10-item version, to be used in the present study, as demonstrating excellent psychometric properties, namely reliability, internal consistency, and construct validity.

SECONDARY OUTCOMES:
Mayo Portland Adaptability Inventory-4 (MPAI-4) | Change from Baseline to Post-Treatment (5 weeks after Baseline)
  The MPAI-4 is comprised of 30 items rated from 0 - 4 with higher scores indicating greater problem severity. Items are subdivided into three subscales reflecting emotional and behavioral self-regulation (Adjustment Index), cognitive and physical abilities (Ability Index), and community integration (Participation Index). T-scores are obtained based on norms derived from a brain injury sample. The present investigation will focus on the former two subscales. Adjustment Index items relate to anxiety, depression, irritability, anger, social interaction, and self-awareness. The Ability Index includes items relating to verbal and nonverbal communication and problem solving ability. Research has provided evidence of good concurrent, construct, and predictive validity as well as satisfactory internal consistency. Sensitivity to treatment-related change has also been substantiated.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Kreutzer, PhD, Principal Investigator — Professor, Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States